CLINICAL TRIAL: NCT07172607
Title: The Effect of Avnace eZZe on Sleep Improvement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202505031
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Sleep Disorder (Disorder); Anxiety Depression Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Avance eZZe (Experimental)
  Interventions: Dietary Supplement: Avance eZZe drink
- Avance eZZe (without liposomal) (Active Comparator)
  Interventions: Dietary Supplement: Avance eZZe drink (without liposomal)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Avance eZZe drink — 25 mL liquid sachet, 1 sachet/day, consume 1 sachet of the sample 1 hour before sleep daily
  Arms: Avance eZZe
Dietary Supplement: Avance eZZe drink (without liposomal) — 25 mL liquid sachet, 1 sachet/day, consume 1 sachet of the sample 1 hour before sleep daily
  Arms: Avance eZZe (without liposomal)
Dietary Supplement: Placebo drink — 25 mL liquid sachet, 1 sachet/day, consume 1 sachet of the sample 1 hour before sleep daily
  Arms: Placebo

SUMMARY:
This study aims to examine the effectiveness of Avance eZZe drink with liposomal technology in improving sleep quality. Participants will be randomly assigned to either the placebo group, Avance eZZe drink group, and Avance eZZe drink without liposomal group, with 25 participants in each group. On the day of the experiment (day 0), participants are required to fill out questionnaires assessing sleep disorders and stress condition, and use a sleep monitoring system to track their sleep and autonomic nervous system conditions. Subsequently, participants will be given the experimental samples and instructed to consume them 1 hour before sleep daily for 28 days. Follow-up assessments will be conducted in the day-1, day-14 and day-28, participants are required to fill out questionnaires assessing sleep disorders and stress condition, and use a sleep monitoring system to track their sleep and autonomic nervous system conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 years or older;
* Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5) criteria for Insomnia Disorder;
* Regular bedtime, between 21:00 and 01:00 and regular wake time;
* Insomnia Severity Index (ISI) score ≥15;
* All medications or interventions for insomnia, mental or physical disorders must have been stable for at least four weeks prior to screening, and participants had to be willing to maintain a stable regimen throughout the study;
* No consumption of sleep or stress-related supplements for at least four weeks prior to screening;
* Willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

* A current diagnosis of sleep-related breathing disorder, periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder;
* Depressive symptoms at screening were considered significantly severe with a PHQ-9 score > 14
* Anxiety symptoms at screening were considered significantly severe with a GAD-7 score > 15;
* Females who are breastfeeding or pregnant;
* Females of childbearing potential who are not practicing acceptable pregnancy prevention methods (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal or have been sterilized surgically.);
* Excessive caffeine use that in the opinion of the investigator contributes to the participant's insomnia, or habitually consumes caffeine-containing beverages after 18:00 and is unwilling to forego caffeine after 18:00 for the duration of his/her participation in the study;
* History of drug or alcohol dependency or abuse within approximately the previous 2 years;
* Current evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal, neurological, or psychiatric disease or malignancy or chronic pain that in the opinion of the investigator could affect the participant's safety or interfere with the study assessments;
* Scheduled for major surgery during the study;
* Participants known to be allergic to any components of the product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep monitoring | Day-0 (baseline), Day-1, Day-14, Day-28
  The difference of electrocardiosignal between two specific points on the body surface will be used to reflect sleep state.
Sleeping quality | Day-0 (baseline), Day-14, Day-28
  The Pittsburgh Sleep Quality Index (PSQI) will be utilized to assess sleeping quality. The minimum value is 0, the maximum value is 42. The higher the score, the worse the outcome.
Insomnia Severity | Day-0 (baseline), Day-14, Day-28
  The Insomnia Severity Index (ISI) will be utilized to assess insomnia severity. The total score ranges from 0 to 28, with higher scores indicating more severe insomnia.

SECONDARY OUTCOMES:
General level of daytime sleepiness | Day-0 (baseline), Day-14, Day-28
  The Epworth Sleepiness Scale (ESS) will be utilized to assess the general level of daytime sleepiness. The total score ranges from 0 to 24, with higher scores indicating greater daytime sleepiness.
Depression severity | Day-0 (baseline), Day-14, Day-28
  Patient Health Questionnaire-9 (PHQ-9) will be utilized to assess depression level. The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms.
Anxiety severity | Day-0 (baseline), Day-14, Day-28
  Generalized Anxiety Disorder-7 (GAD-7) will be utilized to assess anxiety level. The total score ranges from 0 to 21, with higher scores indicating greater anxiety severity.
Low Frequency/High Frequence (LF/HF) ratio | Day-0 (Baseline), Day-1, Day-14, Day-28
  A sleep monitoring system will be utilized to measure LF/HF ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Chien Lee, Doctor, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan